CLINICAL TRIAL: NCT01960374
Title: A Phase I, Single-centre, Open-label, Dose-escalation Study to Assess the Safety, Tolerability and Pharmacokinetics of Selumetinib Given Orally in Japanese and Non-Japanese Asian Healthy Male Volunteers
Brief Title: Dose-escalation Study to Assess Selumetinib Safety, Tolerability and PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: D1532C00086
Record Dates: First submitted 2013-10-09; First posted 2013-10-10 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Healthy Volunteers Pharmacokinetic Study
Keywords: RAS or RAF oncogenes, Inhibition of MEK pathway, inhibition cancer cell proliferation promising anti-cancer therapeutic strategy.
MeSH Terms: interventions — AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Japanese Arm (Experimental): 3 cohorts of 9 subjects. Each cohort will receive oral 25 mg, 50 mg (anticipated) or 75 mg (anticipated) selumetinib (AZD6244; ARRY-142886) (Hyd-Sulfate).
  Interventions: Drug: Selumetinib
- Non-Japanese Asian Arm (Experimental): 3 cohorts of 9 subjects. Each cohort will receive oral 25 mg, 50 mg (anticipated) or 75 mg (anticipated) selumetinib (AZD6244; ARRY-142886) (Hyd-Sulfate).
  Interventions: Drug: Selumetinib

INTERVENTIONS:
Drug: Selumetinib — 1, 2 or 3 x 25 mg selumetinib (AZD6244; ARRY-142886) (Hyd-Sulfate) capsule administered orally as a single dose on Day 1 of the study (total dose 25 mg, 50 mg and 75 mg respectively) with 240 ml of water at room temperature.
  Other Names: (AZD6244; ARRY-142886) (Hyd-Sulfate)

SUMMARY:
The purpose of the study is to assess the safety, tolerability and PK of selumetinib (AZD6244; ARRY-142886) (Hyd-Sulfate) in healthy male Japanese and non-Japanese Asian volunteers following administration of a single dose. Standard safety assessments including ECGs, vital signs, blood/urine safety tests, PK samples and monitoring of adverse events and an optional exploratory pharmacogenetics will be performed.

DETAILED DESCRIPTION:
A Phase I, Single-centre, Open-label, Dose-escalation Study to Assess the Safety, Tolerability and Pharmacokinetics of Selumetinib (AZD6244; ARRY-142886) (Hyd-Sulfate) Given Orally in Japanese and Non-Japanese Asian Healthy Male Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study-specific procedures.
* Non-smokers for at least three months prior to drug administration.
* Healthy male volunteers aged 18 to 55 years with suitable veins for cannulation or repeated venipunctures.
* Subjects included will be either healthy first generation Japanese, or healthy first generation non-Japanese Asian (e.g. Korean, Chinese).
* Japanese subjects must meet the following requirements in order to participate in the study:

  * Subject was born in Japan, Parents and grandparents (both maternal and paternal) are Japanese
  * Subject is in possession of a valid Japanese passport, Expatriate of Japan for not longer than 5 years.
* Non-Japanese Asian subjects must meet the following requirements in order to participate in the study:

  * Subject was born in an Asian country other than Japan, (such as Korea, China, Taiwan etc but not India), Parents and grandparents (both maternal and paternal) are non-Japanese Asian
  * Subject is in possession of a valid passport from their country of origin, Expatriate of their country of origin for not longer than 5 years;
* Have a BMI between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg, inclusive.
* Must use acceptable methods of contraception if the male subject's partner could become pregnant from the time of the first administration of treatment or study medication until 3 months following administration of the last treatment or dose of study medication.

Exclusion Criteria:

* History of any clinically important disease or disorder which, in the opinion of the investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
* Any clinically significant abnormalities in clinical chemistry, haematology, or urinalysis results, as judged by the Investigator.
* Any positive result on screening for serum hepatitis B surface antigen (HbsAg), anti hepatitis core antibody (anti HBc Ig G [and anti HBc IgM if IgG is positive], hepatitis C antibodies (anti HCV), and HIV 1 and 2 antibodies (anti HIV 1/2).
* Abnormal vital signs, after 10 minutes supine rest.
* Current or past history of central serous retinopathy or retinal vein thrombosis, intraocular pressure greater than 21 mmHg or uncontrolled glaucoma.
* Known or suspected history of drug abuse, as judged by the Investigator.
* History of alcohol abuse or excessive intake of alcohol, as judged by the Investigator.
* Positive screen for drugs of abuse or cotinine (nicotine) or positive screen for alcohol at screening or on admission to the study centre on Day -1.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to selumetinib.
* Excessive intake of caffeine-containing drinks or food eg, coffee, tea, chocolate, Red Bull, or cola (more than 6 units of caffeine per day).
* Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IP.
* Use of any prescribed or non prescribed medication including antacids, analgesics other than paracetamol/acetaminophen 1 g 4 times a day for occasional use, herbal remedies, vitamins, and minerals during the 2 weeks or five half-lives of the compound, whichever is longer, prior to the first administration of IP.
* Any intake of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade, or other products containing grapefruit or Seville oranges within 7 days of the first admission on Day -1.Plasma donation within 1 month of screening or any blood donation/blood loss greater than 500 mL during the 3 months prior to screening.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) or has participated in any other clinical study that included drug treatment within at least 3 months of the first administration of IP in this study.
* The period of exclusion begins 3 months after the final dose or 1 month after the last visit whichever is the longest. Note: volunteers consented and screened, but not randomized in this study or a previous Phase I study, are not excluded.Previous administration of study IP in the present study.- involvement in the planning and/or conduct of the study of any RPL/third party contractor or AstraZeneca employee and their close relatives regardless of their role in accordance with their internal procedures.- judged by the Investigator that the volunteer should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.-
* Volunteers who have previously received selumetinib.
* Volunteers who are vegans or have medical dietary restrictions.
* Volunteers who cannot communicate reliably with the Investigator.
* In addition, any of the following is regarded as criteria for exclusion from the genetic research: Previous bone marrow transplant, non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 117 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of selumetinib by assessment of maximum plasma selumetinib concentration (Cmax) | Plasma will be collected at the following time points pre-dose then 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36 and 48 hours post dose
  Rate and extent of absorption of selumetinib following oral doses of selumetinib by assessment of maximum plasma selumetinib concentration (Cmax). Metabolite to parent drug ratios will be calculated for the primary PK parameters AUC and Cmax, and AUC (0-t) if applicable.
Pharmacokinetics of selumetinib by assessment of area under the plasma concentration time curve from zero to infinity (AUC) | Plasma will be collected at the following time points pre-dose then 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36 and 48 hours post dose
  Rate and extent of absorption of selumetinib following oral doses of selumetinib by assessment of area under the plasma concentration time curve from zero to infinity (AUC). Metabolite to parent drug ratios will be calculated for the primary PK parameters AUC and Cmax, and AUC (0-t) if applicable.
Pharmacokinetics of selumetinib by assessment of area under the plasma concentration time curve from zero to the last measurable time point, AUC0-t, if AUC is not adequately measurable | Plasma will be collected at the following time points pre-dose then 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36 and 48 hours post dose
  Rate and extent of absorption of selumetinib following oral doses of selumetinib by assessment of area under the plasma concentration time curve from zero to the last measurable time point, AUC0-t, if AUC is not adequately measurable. Metabolite to parent drug ratios will be calculated for the primary PK parameters AUC and Cmax, and AUC (0-t) if applicable.

SECONDARY OUTCOMES:
Assessment of the Safety and Tolerability of Selumetinib by collection of adverse event reports | All AEs will be collected from Day -1, throughout the treatment periods, and including the follow-up period, assessed after minimum of 7 days. SAEs will be recorded from the time of informed consent.
  Assessment of adverse events (AEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v4.0
Pharmacogenetics | Optional exploratory sample for pharmacogenetics can be taken any time between Day 1 and Day 3 after dosing.
  DNA samples may be used to explore how genetic variations may affect the response to selumetinib. PGx samples will be analysed for BCRP (breast cancer resistance protein), CYP2C19 (cytochrome P450 2C19) and UGT1A1 (UDP glucuronosyltransferase 1A1) genotypes. These transporter and enzymes are known to be polymorphic and maybe involved in the disposition of selumetinib. An assessment of subject's genotype for these transporter/enzymes and subjects PK will be made to see if there is any association of genotype and PK exposure.
Determine safety and tolerability of selumetinib by assessment of 12 lead electrocardiograms | Triplicate 12-lead ECG evaluated at screening & admission. Single 12-lead paper ECGs will follow all dECGs. Digital ECGs will be taken on Day 1 & Day 2 (pre-dose, 1.5h, 2.5h, 4h, 6h, 24h, 48h (pECG only)) & at follow up, at least 7 days after dose.
  Assessment of standard 12 lead electrocardiograms (ECGs)
Determine safety and tolerability of selumetinib by physical examination | At screening and follow up (at least 7 days after dose) full physical examination will be performed. On admission and discharge (day 3) from the CPU a brief physical examination will be performed.
  Assessment of physical examination
Determine safety and tolerability of selumetinib by assessment of vital signs | Supine blood pressure and pulse and oral body temperature will be evaluated at screening and admission, Day 1 (at pre-dose, 1.5h and 6h), Day 2, Day 3 and at follow up at follow up, at least 7 days after dose.
  Assessment of standard vital signs (including blood pressure, pulse)
Determine safety and tolerability of selumetinib by assessment of clinical chemistry results | Clinical chemistry will be evaluated at screening, Day -1, Day 2 and at follow up, at least 7 days after dose.
  Assessment of lab parameters (clinical chemistry)
Determine safety and tolerability of selumetinib by assessment of haematology results | Haematology will be evaluated at screening, Day -1, Day 2 and at follow up, at least 7 days after dose.
  Assessment of lab parameters (haematology)
Determine safety and tolerability of selumetinib by assessment of urinalysis results | Urinalysis results will be evaluated at screening, Day-1 , Day 3 and follow up.
  A sample for urinalysis to be collected along with the other clinical laboratory evaluations. Microscopy should only be performed if the urinalysis result is abnormal.
Determine safety and tolerability of selumetinib by assessment of opthalmic examination | At baseline
  Ophthalmic examination (best corrected visual acuity, IOP and slit-lamp fundoscopy) will be conducted at screening (will be considered the baseline value; no need to repeat) and for cause (on occurrence of AE only).
Pharmacokinetics of selumetinib by assessment of area under the plasma concentration time curve from zero to the last measurable time point, AUC0-t. | Plasma will be collected at the following time points pre-dose then 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36 and 48 hours post dose
  Rate and extent of absorption of selumetinib following oral doses of selumetinib by assessment of area under the plasma concentration time curve from zero to the last measurable time point, AUC0-t. Metabolite to parent drug ratios will be calculated for the primary PK parameters AUC and Cmax, and AUC (0-t) if applicable.
Pharmacokinetics of selumetinib by assessment of area under the plasma concentration time curve from zero to 12h time point, AUC0-12. | Plasma will be collected at the following time points pre-dose then 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36 and 48 hours post dose
  Rate and extent of absorption of selumetinib following oral doses of selumetinib by assessment of area under the plasma concentration time curve from zero to 12h time point, AUC0-12. Metabolite to parent drug ratios will be calculated for the primary PK parameters AUC and Cmax, and AUC (0-t) if applicable.
Pharmacokinetics of selumetinib by assessment of area under the plasma concentration time curve from zero to 24h time point, AUC0-24. | Plasma will be collected at the following time points pre-dose then 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36 and 48 hours post dose
  Rate and extent of absorption of selumetinib following oral doses of selumetinib by assessment of area under the plasma concentration time curve from zero to 24h time point, AUC0-24. Metabolite to parent drug ratios will be calculated for the primary PK parameters AUC and Cmax, and AUC (0-t) if applicable.
Pharmacokinetics of selumetinib by assessment of time to reach maximum plasma concentration for selumetinib (tmax). | Plasma will be collected at the following time points pre-dose then 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36 and 48 hours post dose
  Rate and extent of absorption of selumetinib following oral doses of selumetinib by assessment of time to reach maximum plasma concentration for selumetinib (tmax).
Pharmacokinetics of selumetinib by assessment of selumetinib apparent clearance (CL/F). | Plasma will be collected at the following time points pre-dose then 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36 and 48 hours post dose
  Rate and extent of absorption of selumetinib following oral doses of selumetinib by assessment of of selumetinib apparent clearance (CL/F).
Pharmacokinetics of selumetinib by assessment of rate of the elimination half-life of selumetinib from circulation following single oral dose (t½). | Plasma will be collected at the following time points pre-dose then 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36 and 48 hours post dose
  Rate and extent of absorption of selumetinib following oral doses of selumetinib by assessment of rate of the elimination half-life of selumetinib from circulation following single oral dose (t½).
Pharmacokinetics of selumetinib by assessment of volume of distribution divided by bioavailability (Vss/F; estimate of steady state distribution volume for selumetinib following single oral dose). | Plasma will be collected at the following time points pre-dose then 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36 and 48 hours post dose
  Rate and extent of absorption of selumetinib following oral doses of selumetinib by assessment of volume of distribution divided by bioavailability (Vss/F; estimate of steady state distribution volume for selumetinib following single oral dose).

CONTACTS AND LOCATIONS:
Overall Officials: Ian C Smith, MD, Study Chair — AstraZeneca UK, MSD; Ulrike Lorch, MD, Principal Investigator — Richmond Pharmacology Ltd, UK
Locations (1):
- Research Site, London, United Kingdom